CLINICAL TRIAL: NCT02554357
Title: Quality of Analgesia After Interscalene Block With Bupivacaine and Exparel® vs. Bupivacaine Alone After Arthroscopic Shoulder Surgery
Brief Title: Quality of Analgesia After Interscalene Block After Arthroscopic Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North American Institute for Continuing Medical Education (NAICE) (Other)
Collaborators: New York School of Regional Anesthesia (Other); Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NAICE-002
Record Dates: First submitted 2015-07-11; First posted 2015-09-18 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Injury of Shoulder Region
MeSH Terms: conditions — Shoulder Injuries | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exparel block in arthroscopic surgery (Experimental): Evaluation of Exparel block in arthroscopic shoulder surgery.
  Interventions: Drug: Exparel block in arthroscopic shoulder surgery
- Bupivacaine block in shoulder surgery (Experimental): Evaluation of Bupivacaine block in shoulder surgery.
  Interventions: Drug: Bupivacaine block in shoulder surgery

INTERVENTIONS:
Drug: Exparel block in arthroscopic shoulder surgery — The interscalene block will be performed with ultrasound guidance and nerve stimulation.
  Other Names: ISBPB with bupivacaine and Exparel
  Arms: Exparel block in arthroscopic surgery
Drug: Bupivacaine block in shoulder surgery — The interscalene block will be performed with ultrasound guidance and nerve stimulation.
  Other Names: ISBPB with bupivacaine alone
  Arms: Bupivacaine block in shoulder surgery

SUMMARY:
Shoulder arthroscopic causes post operative pain that outlasts analgesia provided by single injection nerve blocks.

DETAILED DESCRIPTION:
The interscalene brachial plexus block (ISBPB) is a common analgesic technique for procedures of the shoulder and upper arm.

Moreover, the incidence of rebound pain is well documented and is often of considerable discomfort to patients, who may quickly go from little or no pain to moderate-severe pain. Continuous nerve block techniques with home ambulatory catheters are currently utilized to manage postoperative pain.This study is designed to compare the level and duration of pain control of Exparel® injected after bupivacaine via stop-cock connected syringes and bupivacaine alone for ISBPB.

ELIGIBILITY:
Inclusion Criteria:

* Dutch or English speaking adults
* 18 years or older ASA I-III physical class
* Scheduled for elective arthroscopic shoulder surgery

Exclusion Criteria:

* History of allergy to a local anesthetic
* Baseline neurological deficit
* Medical condition that would make it difficult to assess sensory distribution or communicate with the investigators' staff
* Recent history (< 3 months) of drug or alcohol abuse
* Concomitant opioid therapy
* Preexisting coagulation disorder
* Infection at the injection site
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Worst pain | assessed by the Modified Brief Pain Inventory short form Question 1 in the first postoperative week - postoperative day (POD) 1 through POD7
Satisfaction with analgesia | assessed by the Overall Benefit of Analgesia Score (OBAS) in the first postoperative week postoperative day (POD)1 through POD7

SECONDARY OUTCOMES:
Onset of sensory block | onset will be measured up to 30 minutes
Duration of sensory block | duration will be measured up to 72 hours
Onset of motor block | onset will be measured up to 30 minutes
duration of motor block | duration will be measured up to 72 hours
functionality of the surgical arm | assessed on the scale 0-5 in the first postoperative week - postoperative day (POD) 2- POD7

CONTACTS AND LOCATIONS:
Overall Officials: Admir Hadzic, MD, Study Director — Director
Locations (2):
- Belgium (2):
  - Department of Anesthesiology Ziekenhuis Oost-Limburg, Genk
  - Department of Anesthesiology ZOL, Genk

REFERENCES:
- [Derived] Vandepitte C, Kuroda M, Witvrouw R, Anne L, Bellemans J, Corten K, Vanelderen P, Mesotten D, Leunen I, Heylen M, Van Boxstael S, Golebiewski M, Van de Velde M, Knezevic NN, Hadzic A. Addition of Liposome Bupivacaine to Bupivacaine HCl Versus Bupivacaine HCl Alone for Interscalene Brachial Plexus Block in Patients Having Major Shoulder Surgery. Reg Anesth Pain Med. 2017 May/Jun;42(3):334-341. doi: 10.1097/AAP.0000000000000560. PMID 28157791